CLINICAL TRIAL: NCT05763550
Title: A Multicenter, Randomized, Double-Blind, Double-Dummy , Pregaballin-Controlled, Phase 2 Study to Evaluate the Efficacy and Safety of HSK16149 Capsules in Chinese Patients With Herpetic Neuralgia
Brief Title: To Evaluate the Efficacy and Safety of HSK16149 Capsule in Chinese Patients With Herpetic Neuralgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSK16149-205
Record Dates: First submitted 2023-02-28; First posted 2023-03-10 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-02

CONDITIONS: Herpetic Neuralgia
MeSH Terms: interventions — BID protein, human; Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HSK16149 20mg BID (Experimental)
  Interventions: Drug: HSK16149 20mg BID
- HSK16149 40mg BID (Experimental)
  Interventions: Drug: HSK16149 40mg BID
- Pregabalin 150mg BID (Active Comparator)
  Interventions: Drug: Pregabalin 150mg

INTERVENTIONS:
Drug: HSK16149 20mg BID — HSK16149 20mg, orally twice a day, treatment period; 4-weeks fixed dose.
  Arms: HSK16149 20mg BID
Drug: HSK16149 40mg BID — HSK16149 40mg, orally twice a day, treatment period; 4-weeks fixed dose.
  Arms: HSK16149 40mg BID
Drug: Pregabalin 150mg — pregabalin, orally twice a day, treatment period; 150 mg (75 mg twice daily) for 1 week；300 mg (150 mg twice daily) daily for 3 week
  Arms: Pregabalin 150mg BID

SUMMARY:
Investigate the efficacy and safety of HSK16149 capsules in Chinese herpetic Neuralgia following 4 weeks treatment in comparison to pregabalin.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent;
* Males or females aged 18 years and older ;
* Patients must have herpetic neuralgia;
* At Screening, pain scale (VAS) of ≥ 40 mm;
* At Screening, pain scale (NRS) of ≥ 4.

Exclusion Criteria:

* Patients have pain present for more than 1 months after the healing of the herpes zoster skin rash;
* AST/ALT > 2 × upper limit of normal (ULN), or TBIL≥1.5 × ULN;
* Serum Creatine > 176μmol/L;
* Any active infections at screening;
* History of allergic or medically significant adverse reaction to investigational products or their excipients, pregabalin or related compounds;
* Participated in another clinical study within 30 days prior to screening;
* Pregnant or breastfeeding at screening ;
* Other conditions unlikely to participate in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-08-07 (Actual)

PRIMARY OUTCOMES:
Compare the change from baseline in Numeric Rating Scales(NRS )between HSK16149 and pregabalin at week 4 | Baseline and week 4
  Numeric Rating Scales(NRS )was a 11-point numeric rating scale ( 0[no pain] to 10 [worst possible pain]

SECONDARY OUTCOMES:
Compare the response rate between HSK16149 and pregabalin at week 4 (Proportion of subjects whose NRS decreased by ≥30% and≥ 50% from baseline ) | Baseline and week 4
Compare the change from baseline in VAS between HSK16149 and pregabalin at week 4 | Baseline and week 4
  VAS, in which the participant rates pain on a 100 mm-long horizontal line, where 0 mm = no pain and 100 mm = worst possible pain
Compare the change from baseline in DSIS between HSK16149 and pregabalin at week 4 | Baseline and week 4
  The sleep interference scores on a scale of 0-10, where 0 = pain did not interfere with sleep to 10 = pain completely interfered with sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Fangqiong Li, Study Chair — Haisco
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China